CLINICAL TRIAL: NCT06290375
Title: A Multi-center Stage II Trial to Evaluate the Efficacy, Safety, and Pharmacokinetic Profile of HSK21542 Tablets for the Treatment of Moderate-to-severe Pruritus in Peritoneal Dialysis Subjects
Brief Title: A Study of HSK21542 in a Peritoneal Dialysis Pruritus Population.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xizang Haisco Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK21542-T-202
Record Dates: First submitted 2024-02-07; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Pruritus
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK21542 tablet 2mg (Experimental)
  Interventions: Drug: HSK21542 tablet
- Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK21542 tablet — once-daily
  Arms: HSK21542 tablet 2mg
Drug: Placebo — once-daily
  Arms: Placebo

SUMMARY:
This is a two- stage study. Stage I is a multicenter, open-label trial；Stage II was a multi-center, randomized, double-blind, placebo-controlled trial. About 250 maintenance peritoneal dialysis patients with moderate or above pruritus are planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 and ≤ 75 years old, male or female;
2. Dry weight at screening: 40.0-135.0 kg (inclusive);
3. Patients who have received regular peritoneal dialysis for at least 3 months prior to screening；
4. Male subjects who agree to use condoms in sexual intercourse during the study and within 3 months after the last dose; female subjects who have been menopausal for at least one year, or who have been sterilized permanently (e.g., fallopian tube occlusion, hysterectomy, bilateral salpingectomy); or women of childbearing potential who agree to take effective contraceptive measures during the study and within 3 months after the last dose, such as oral contraceptives, condoms, and contraceptive films；
5. Subjects who are willing to sign an informed consent form, fully understand the objectives and significance of the trial, and are willing to comply with the trial protocol before any of the study-related procedures start.

Exclusion Criteria:

1. Having a history of allergy to opioids, such as urticaria ；
2. Expecting to undergo hematodialysis and/or renal transplantation during the study；
3. Expecting to undergo parathyroidectomy during the study；
4. Pruritus that not be caused by CKD or its complications ；
5. New or change of treatment received for peritoneal dialysis within 3 months prior to screening or anticipating to adjust peritoneal dialysis during the study
6. Subjects must not have any of the following medical conditions：

   1. Cerebrovascular accident, myocardial infarction, coronary stent implantation, severe systolic or diastolic heart failure (e.g., congestive heart failure in NYHA class III or higher) within the previous 6 months；
   2. Uncontrolled hypertension at screening was defined as systolic blood pressure >160mmHg or diastolic blood pressure >100mmHg；
   3. Severe mental illness or cognitive impairment (e.g., dementia)；
   4. Any other relevant acute or chronic neurological or psychiatric condition within 3 months prior to screening that, at the discretion of the investigator, is not suitable for enrollment (e.g., encephalopathy, coma, delirium)；
   5. Patients with malignancy, but excluding: curable cervical carcinoma in situ, skin basal cell or squamous cell carcinoma, or any other tumors that have been cured (no evidence of disease recurrence within 5 years)；
   6. Severe uncontrolled infections at screening, including severe abdominal infection, upper respiratory tract infection, lower respiratory tract infection, urinary tract infection, etc；
   7. Inability to understand and complete the scale assessments required by the study protocol。
7. At the screening or baseline, participants have laboratory values that met the following criteria：

   1. Alanine transaminase (ALT) or AST (aspartate transaminase) > 2.5 × upper limit of normal (ULN), or total bilirubin > 2 × ULN at screening；
   2. Blood sodium > 155 mmol/L at screening；
   3. Hemoglobin < 80 g/L at screening；
8. New or change of medications that may affect the judgment of antipruritic efficacy, including but not limited to antipsychotics, sedative-hypnotics, selective serotonin reuptake inhibitors (SSRIs), anxiolytics, or tricyclic antidepressants within 14 days prior to screening or anticipating inevitable treatment regimen adjustment during the study；
9. New or change of treatment received including antihistamines (except for otic or ophthalmic preparations), systemic or topical corticosteroids (except for otic or ophthalmic preparations),calcineurin inhibitors , gabapentin or pregabalin within 7 days prior to screening or anticipating inevitable treatment regimen adjustment during the study;
10. Subjects were receiving UV treatment or were expected to receive this treatment during the trial；
11. Having used opioids within 7 days before screening, or being unable to avoid the use of opioids other than the investigational drug during the study；
12. A history of substance abuse, drug use, and/or alcohol abuse, defined as drinking an average of >2 units of alcohol per day within 3 months prior to screening (1 unit =360mL of 5% beer or 45mL of 40% liquor or 150mL of wine)；
13. Having participated in any clinical trial of other drug or medical device within 1 month before screening (received study medication or treated by the medical device in the clinical trial)；
14. Positive for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), syphilis antibody, or human immunodeficiency virus (HIV) antibody at screening；
15. Females who are pregnant or breastfeeding；
16. Subjects with any other factors considered by the investigator to be ineligible for participation in this clinical study。

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-03-08 (Estimated); Primary Completion 2024-03-08 (Estimated); Study Completion 2025-04-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with an improvement of ≥ 4points from baseline in the weekly average of the daily Worst Itch Numeric Rating Scale (WI-NRS) after 12 weeks of treatment. | Week 12
  In the NRS score, 0-10 represents different degrees of itching, the larger the number, the more severe the itching

SECONDARY OUTCOMES:
Change from baseline in subjects' quality of life (evaluated using the Skindex-10 scale ) after 12 weeks of treatment. | Week 2、4、8、12
  The Skindex-10 Scale is a multidimensional questionnaire which assesses itch-related quality of life over the past week. The questions cover 3 domains: symptoms, emotions, and functioning domain. A lower total score represents better quality of life.
Change from baseline in subjects' quality of life (evaluated using the 5-D itch scale) after 12 weeks of treatment. | Week 2、4、8、12
  The 5-D Itch Scale is a multidimensional questionnaire which assesses itch-related quality of life over the past 2 weeks. The questions cover five dimensions of itch including the degree, duration of itch/day, direction (improvement/worsening), disability (impact on activities such as work), and body distribution of itch. A lower total score represents better quality of life